CLINICAL TRIAL: NCT03457948
Title: A Pilot Study of Pembrolizumab and Liver-Directed Therapy or Peptide Receptor Radionuclide Therapy for Patients With Well-Differentiated Neuroendocrine Tumors and Symptomatic and/or Progressive Metastases
Brief Title: Pembrolizumab With Liver-Directed or Peptide Receptor Radionuclide Therapy for Neuroendocrine Tumors and Liver Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nicholas Fidelman, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); BTG International Inc. (Other)
Responsible Party: Sponsor-Investigator, Nicholas Fidelman, MD, Assistant Professor of Clinical Radiology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17705; NCI-2018-00227 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2018-02-27; First posted 2018-03-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Malignant Neoplasm in the Liver; Neuroendocrine Neoplasm
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — pembrolizumab; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group I [pembrolizumab, 177Lu DOTATATE] (Experimental): Patients will be treated with pembrolizumab and intravenous peptide receptor radionuclide therapy (PRRT) using 177Lu-DOTA0-Tyr3-Octreotate (177Lu-DOTATATE, Lutathera®) for up to four (4) sessions. Patients with somatostatin receptor positive (SSTR+) tumors with Ki-67 index > 20% (well-differentiated grade 3) and any number of liver and/or extrahepatic lesions with liver parenchyma replacement by tumor < 75%. Patients who achieve progressive or stable disease response after cycle 4 may receive an additional 4 cycles of pembrolizumab and lutetium Lu-177 DOTATATE in the absence of disease progression or unacceptable toxicity and pembrolizumab for up to 35 cycles.
  Interventions: Biological: Pembrolizumab; Biological: Peptide Receptor Radionuclide Therapy (PRRT) using 177Lu-DOTA0-Tyr3-Octreotate
- Group II [pembrolizumab, TAE] (CLOSED) (Experimental): Patients receive pembrolizumab as in Group I. Patients with any number of liver lesions, largest being no larger than 5 cm, who have < 75% liver parenchyma replacement by tumors, undergo Arterial Embolization (TAE) over 2-3 hours, 3-7 days following the first dose of pembrolizumab.
  Interventions: Procedure: Arterial Embolization; Biological: Pembrolizumab
- Group III [pembrolizumab, yttrium-90 microsphere RE] (CLOSED) (Experimental): Patients receive pembrolizumab as in Group I. Patients with any number of liver lesions, largest measuring more than 5 cm, who have < 75% liver parenchyma replacement by tumors, undergo yttrium-90 microsphere Radio Embolization (RE) 3-15 days following the first dose of pembrolizumab.
  Interventions: Biological: Pembrolizumab; Device: Yttrium-90 Microsphere Radioembolization

INTERVENTIONS:
Procedure: Arterial Embolization — Undergo TAE
  Other Names: TAE; Transarterial Embolization
  Arms: Group II [pembrolizumab, TAE] (CLOSED)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Peptide Receptor Radionuclide Therapy (PRRT) using 177Lu-DOTA0-Tyr3-Octreotate — Given IV
  Other Names: Lutathera; 177Lu-DOTATATE
  Arms: Group I [pembrolizumab, 177Lu DOTATATE]
Device: Yttrium-90 Microsphere Radioembolization — Undergo yttrium-90 microsphere RE
  Other Names: Yttrium Y 90 Microsphere Therapy; Yttrium-90 Radioembolization; Yttrium-90 Microsphere RE
  Arms: Group III [pembrolizumab, yttrium-90 microsphere RE] (CLOSED)

SUMMARY:
This pilot phase II trial studies how effective pembrolizumab and liver-directed therapy or peptide receptor radionuclide therapy are at treating patients with well-differentiated neuroendocrine tumors and symptomatic and/or progressive tumors that have spread to the liver (liver metastases). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Liver-directed therapies such as radiofrequency ablation, transarterial embolization, yttrium-90 microsphere radioembolization, and cryoablation may help activate the immune system in order to shrink tumors that are not being directly targeted. Peptide receptor radionuclide therapy is a form of targeted treatment that is performed by the use of a small molecule, which carries a radioactive component attached to a peptide. Once injected into the body, this small molecule binds to some specific sites on tumor cells called receptors and emit medium energy radiation that can destroy cells. Because this radionuclide is attached to the peptide, which binds receptors on tumor lesions, the radiation can preferably be targeted to the tumor cells in order to destroy them. Giving pembrolizumab in combination with liver-directed therapy or peptide receptor radionuclide therapy may work better than pembrolizumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate safety profile of pembrolizumab in combination with Peptide Receptor Radionuclide Therapy (PRRT), transarterial embolization, and radioembolization.

II. To evaluate the best observed overall response rate (ORR) in lesion(s) not targeted for liver-directed therapy (abscopal effect) to pembrolizumab plus liver-directed therapy according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for patients with metastatic well-differentiated (WD) neuroendocrine tumors (NET)s (WD-NETs).

III. To evaluate the best observed ORR to pembrolizumab plus peptide receptor radionuclide therapy (PRRT) according to RECIST 1.1 for patients with metastatic grade 2 and 3 WD-NET (Ki-67 > 10%).

SECONDARY OBJECTIVES:

I. To evaluate duration of response (DOR) in patients receiving pembrolizumab in combination with liver-directed therapies or PRRT.

II. To evaluate progression free survival (PFS) in subjects treated with pembrolizumab in combination with liver-directed therapies or PRRT.

III. Best observed radiographic ORR per modified RECIST (mRECIST) in lesions targeted for liver-directed therapy.

IV. Duration of response in lesions targeted for liver-directed therapy by mRECIST.

EXPLORATORY OBJECTIVES:

I. To compare ORR, DOR, and PFS based on immune-related (ir)RECIST with the same measures assessed by RECIST 1.1.

II. To correlate clinical outcomes (ORR, DOR, PFS) with baseline immune cell infiltration and PD-L1 staining in cycle 1 and cycle 5 tumor biopsies.

III. To assess the level of PD-L1 expression in tumor tissue prior to liver-directed therapy (prior to PRRT) and 5 weeks following liver-directed therapy (following PRRT).

IV. To assess T cell infiltration on the pre-177Lu-DOTATATE (pre-PRRT) and on the on-treatment tumor tissue biopsies.

V. To assess baseline circulating T cell receptor (TCR) repertories and changes in TCR repertories with treatment, and correlate baseline and turnover of repertories to clinical outcomes.

VI. To analyze the relationship between baseline tumor proliferative index (as measured by Ki67) and response to therapy.

OUTLINE: Patients originally assigned to 1 of 3 groups. As of 09/15/2022, Groups 2 and 3 are closed to enrollment.

GROUP I (PRRT): Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity. PRRT using 177Lu-DOTATATE(Lutathera®) will be offered to patients with somatostatin receptor positive (SSTR+) tumors with Ki-67 index > 20% (well-differentiated grade 3). Patients may have any number of liver and/or extrahepatic lesions with liver parenchyma replacement by tumor < 75%. 200±20 millicurie (mCi) of 177Lu-DOTATATE will be administered intravenously per treatment on outpatient basis. Patients will receive a total of four treatments of 177Lu-DOTATATE, administered every 8±1 weeks. Patients with partial response (PR) or stable disease (SD) by RECIST v. 1.1 after cycle 4 of pembrolizumab who were treated with PRRT (group 1) would continue to receive systemic IV administrations of 177Lu-DOTATATE every 8 +/-1 weeks for up to four (4) treatments. After completion of four (4) PRRT treatments, pembrolizumab may be administered alone for up to 35 cycles

CLOSED - GROUP II (TRANSARTERIAL EMBOLIZATION (TAE)): Patients receive pembrolizumab as in Group I. Patients with any number of liver lesions, largest being no larger than 5 cm, who have < 75% liver parenchyma replacement by tumors, undergo TAE over 2-3 hours, 3-7 days following the first dose of pembrolizumab.

CLOSED - GROUP III (RADIOEMBOLIZATION (RE)): Patients receive pembrolizumab as in Group I. Patients with any number of liver lesions, largest measuring more than 5 cm, who have < 75% liver parenchyma replacement by tumors, undergo yttrium-90 microsphere RE 3-15 days following the first dose of pembrolizumab.

After completion of study treatment, patients are followed up at 30 days and then every 3-6 months thereafter.

ELIGIBILITY:
Subject Inclusion Criteria

1. Be willing and able to provide written informed consent for the trial.
2. Be >= 18 years of age on day of signing informed consent.
3. Have a histologically proven well-differentiated neuroendocrine tumor (WHO grade 1, grade 2, or morphologically and/or clinically well-differentiated grade 3) of any primary site, including unknown primary site.

   a. For group 1, only well-differentiated grade 2 or 3 tumors with Ki-67 index > 10% that demonstrate somatostatin receptor expression on DOTA or In-111 Octreoscans will be allowed.
4. Radiographic, biochemical, or clinical evidence of tumor progression over a period of up to 12 months in at least one site.

   1. Group 1: At least one symptomatic and/or progressive somatostatin receptor positive (SSTR+) lesion over a period of up to 12 months, or have at least one measurable lesion based on RECIST v. 1.1.
   2. Groups 2-3: At least one symptomatic and/or progressive liver lesion over a period of up to 12 months, or have at least two measurable lesions in the liver or at least one measurable lesion in the liver and another measurable lesion elsewhere, based on RECIST v. 1.1.
5. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
6. Have a life expectancy of greater than 3 months.
7. Demonstrate adequate organ function.

   1. Absolute neutrophil count (ANC) >=1,500 /microliters (mcL).
   2. Platelet count >75,000/mcL.
   3. Hemoglobin > 9 g/dL (For group 1 only. There is no hemoglobin cut-off level for groups 2-3).
   4. Serum creatinine OR Measured or calculated a creatinine clearance (GFR can also be used in place of creatinine or CrCl) <=1.5 X upper limit of normal (ULN) OR >=60 mL/min for subject with creatinine levels > 1.5 X institutional ULN.
   5. Serum total bilirubin <= 1.5 X ULN OR Direct bilirubin <= ULN for subjects with total bilirubin levels > 1.5 ULN.
   6. AST (SGOT) and ALT (SGPT) <= 5 X ULN.
   7. Albumin >= 2.5 mg/dL.
   8. International Normalized Ratio (INR) or Prothrombin Time (PT) <=1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thrombin time (PTT) is within therapeutic range of intended use of anticoagulants.
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 30 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Subject Exclusion Criteria

1. Has had prior thermal ablation, embolotherapy, radioembolization, or external beam radiation within 30 days of initiation of study therapy.
2. Has had prior peptide receptor radionuclide therapy (group 1 only).
3. Has had biliary tract intervention that resulted in compromise to the Ampulla of Vater or a biliary-enteric anastomosis (groups 2-3 only).
4. Has greater than 75% liver parenchyma replacement by tumor (determined by radiologist investigator).
5. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
6. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
7. Has a known history of active Tuberculosis (TB) (Bacillus Tuberculosis).
8. Hypersensitivity to pembrolizumab or any of its excipients.
9. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., <=Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
10. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., <=Grade 1 or at baseline) from adverse events due to a previously administered agent.

    1. Note: Subjects with <= Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
    2. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
    3. Concurrent somatostatin analog therapy is allowed.
11. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
12. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease.
15. Has an active infection requiring systemic therapy.
16. Has liver fibrosis either determined by imaging or laboratory testing (i.e. total serum bilirubin > 1.5 times ULN, Aspartate Aminotransferase (AST) and alanine aminotransferase (ALT) > 5 times ULN, INR >1.5 times ULN, albumin <2.0mg/dl).
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
20. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
21. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
22. Has known active untreated Hepatitis B.
23. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with an overall response | At 12 weeks
  The All Subjects as Treated (ASaT, ITT) population will be used for the analysis of ORR. The primary efficacy endpoint will be best observed Overall Response Rate (ORR) by RECIST 1.1 (investigator reported). ORR is defined as the proportion of the subjects in the analysis population who have a complete response (CR) or partial response (PR). The point estimate and 95% confidence interval of overall response rate will be obtained for each of the three groups separately.
Number of treatment-related adverse events (Group 1) | Up to 30 days after the end of treatment
  Adverse events occurring from the start of treatment until 30 days after the end of treatment will be summarized by maximum toxicity grade. All treatment related adverse events will be graded using NCI CTCAE v5.0. Safety analysis will include a tabulation of all toxicities by grade. The frequency of toxicities will be tabulated separately for each cohort.

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 3 years
  Kaplan-Meier method will be used to summarize DOR for participants with a documented complete response or partial response per RECIST v.1.1 criteria. . Median DOR and its 95% confidence interval will be obtained for each of the three liver-directed therapies and PRRT groups separately.
Number of treatment-related adverse events (Groups 2 & 3) | Up to 30 days after the end of treatment
  Adverse events occurring from the start of treatment until 30 days after the end of treatment will be summarized by maximum toxicity grade. All treatment related adverse events will be graded using NCI CTCAE v5.0. Safety analysis will include a tabulation of all toxicities by grade. The frequency of toxicities will be tabulated separately for each cohort.
Median Progression free survival (PFS) | Up to 3 years
  Progression free survival is defined as the time from the first day of study treatment with protocol therapy to the date of documented tumor progression or death due to any cause, whichever occurs first, as determined by RECIST v1.1. Kaplan-Meier methods will be used to estimate PFS with 95% confidence interval for each group separately.
Immune-related progression free survival (irPFS) | Up to 3 years
  Immune-related progression free survival is defined as the time from the first day of study treatment with protocol therapy to the date of documented tumor progression or death due to any cause, whichever occurs first, as determined by immune-related-RECIST (irRC). Kaplan-Meier methods will be used to estimate irPFS with 95% confidence interval for each group separately.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Fidelman, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No